CLINICAL TRIAL: NCT04751149
Title: Acute Urinary Retention After Early, Medium or Late Removal of the Urinary Catheter in Rectal Cancer Surgery. RAOREC Study
Brief Title: Incidence of Acute Urine Retention: Randomized Clinical Trial Comparing Early, Mid or Late Urinary Catheter Removal in Patients With Rectal Resection
Acronym: RAOREC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Donostia (Other)
Responsible Party: Principal Investigator, Prof. Jose M Enríquez-Navascués, PhD; Head of service, Hospital Donostia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ELO-RAO-2019-01
Record Dates: First submitted 2020-10-27; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Rectal Cancer; Retention, Urinary; Urinary Tract Infections; Surgical Site Infection; Anastomotic Leak
MeSH Terms: conditions — Rectal Neoplasms; Urinary Retention; Urinary Tract Infections; Surgical Wound Infection; Anastomotic Leak

STUDY DESIGN:
Intervention Model Description: Early removal of urinary catheter Medial removal of urinary catheter Late removal of urinary catheter
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early Urinary Catheter Removal (Experimental): Urinary Catheter will be removed the first postoperative day after rectal resection
  Interventions: Procedure: Removal of Urinary Catheter
- Medium Urinary Catheter Removal (Experimental): Urinary Catheter will be removed the third postoperative day after rectal resection
  Interventions: Procedure: Removal of Urinary Catheter
- Late Urinary Catheter Removal (Experimental): Urinary Catheter will be removed the fifth postoperative day after rectal resection
  Interventions: Procedure: Removal of Urinary Catheter

INTERVENTIONS:
Procedure: Removal of Urinary Catheter — Urinary catheter will be removed in aeseptic conditions. Before the removal a urinary culture will be obtained from the catheter.

SUMMARY:
DESIGN:

Randomized, open-label and parallel clinical trial, assigned to early, mid, or late withdrawal of urinary catheter with a 1: 1: 1 allocation ratio.

POPULATION:

Patients undergoing anterior rectal resection, low rectal resection, or abdominoperineal amputation for any reason.

OBJECTIVES:

The main objective is to compare the incidence of acute urine retention after removal of the urinary catheter in the postoperative period of rectal resection.

Secondary objectives are:

1. Incidence of urinary tract infection after urinary catheter removal.
2. Incidence of specific postoperative complications (Surgical wound infection, Respiratory infection, Anastomotic dehiscence, ileus).
3. Incidence of postoperative complications assessed according to the Comprehensive Complication Index (CCI) scale.

DESCRIPTION OF THE INTERVENTION:

In all patients, a Rectal Resection (anterior rectal resection, posterior pelvic exenteration or abdominoperineal amputation) will be performed. In group 1A, the urinary catheter will be removed on the 1st postoperative day. In group 1B patients, the urinary catheter will be removed on the 3rd postoperative day. In group 1C patients, the urinary catheter will be removed on the 5th postoperative day. All patients will have a urine culture taken at the time of withdrawal.

DETAILED DESCRIPTION:
Currently there is a trend towards prolonged urinary catheterization in patients undergoing rectal resection surgery. However, there are studies that defend although there is a slight increase in AUR in these patients, it can be withdrawn early in a safe way with a lower incidence of UTI.

The aim of the study is to analyse whether there are differences in the incidence of AUR in rectal surgery patients and to observe whether it has an impact on other postoperative complications. A randomized clinical trial is proposed to compare an early, mid or late removal of the urinary catheter in patients with rectal resection.

- Potential Risks and Benefits:

Both techniques, both early and late withdrawal, are approved practices that are carried out in a standardized way in the current practice. There are no potential risks associated with the study intervention, beyond the intrinsic risks of the procedure itself.

- Objectives of the study:

Main objective: to compare the incidence of acute urine retention after removal of the urinary catheter in the postoperative period of rectal resection.

Secondary objectives:

Incidence of urinary tract infection after urinary catheter removal. Incidence of specific postoperative complications (surgical wound infection, respiratory infection, anastomotic dehiscence, ileus).

Incidence of postoperative complications assessed according to the Comprehensive Complication Index (CCI) scale.

* Variables:

  * Demographic: sex, date of birth, BMI, ASA, Benign Prostate Hyperplasia, surgical history, usual treatment, date of diagnosis of the tumor, neoadjuvant treatment, tumor stage (TNM).
  * Preoperative evaluation: IPSS (International Prostate Syndrome Score) for evaluation of preoperative urinary function in men.
  * Surgical treatment: date of surgery, antibiotic prophylaxis, type of surgical approach, blood volume administered during surgery, mechanical preparation of the colon, type of surgery, ligation of the inferior mesenteric artery (IMA), need for intraoperative transfusion, duration of intervention, bleeding, intraoperative complications.
  * Postoperative evolution: Acute retention of urine, urinary tract infection, surgical wound infection, respiratory infection, paralytic ileus, blood volume administered postoperatively, postoperative complications (ICC), date of diagnosis, reoperation, hospital stay, postoperative mortality and readmission .
  * Evolution and follow-up: Need for catheterization, removal of urinary catheter, urinary tract infection.
* Definitions:
* Postoperative morbidity includes all postoperative complications that occurred during the first 30 postoperative days. Complications will be evaluated according to the CCI (classification that considers the accumulation of complications based on the Clavien-Dindo scale).
* Severe prostate symptomatology is considered to be an IPSS score (established questionnaire for prostate symptoms) greater than 20.
* Urinary catheter placement is considered to be the placement of a catheter through the urethra, always performed under antiseptic conditions.
* AUR is considered the impossibility of urine output despite urinary desire and at least 30 minutes, or anuria of 8 hours after the removal of the UC with a retention of more than 250 mL.
* UTI is defined as a positive urine culture with> 10 5 bacterial colonies / mL of urine.
* Respiratory infection is considered a positive sputum culture and / or a chest radiograph with parenchymal condensations.
* The wound infection is considered deep, superficial or parastomal according to the CDC (Center for Disease Control) criteria for wound infections.
* A delay in oral tolerance due to vomiting, abdominal distention or the need for nasogastric tube placement will be considered ileus.
* Anastomotic dehiscence and its severity is defined according to the International Study Group of Rectal Cancer.
* Postoperative mortality is defined as death within the first 90 days after surgery or before hospital discharge.
* Readmission is defined as admission to the hospital within 30 days of discharge from the hospital.
* Neoadjuvant chemotherapy is considered to be that received prior to surgery.
* The duration of the surgical intervention is considered the time from the beginning of the skin section to the end of the last skin point, calculated in minutes.
* The volume administered during the surgery is considered the volume of fluids administered by the venous route from the induction of anesthesia to the extubation of the patient.
* A high ligation of the IMA is considered to be the ligation that is performed about 2 cm from the root of the IMA, preserving the superior hypogastric plexus. Low ligation of the IMA is considered one that is distal to the bifurcation of the IMA.
* Study Design:

  * Randomized clinical trial, with an allocation ratio of 1: 1: 1, controlled, of patients undergoing rectal resection surgery.
  * The study population is hospitalized patients, who underwent anterior rectal resection, low anterior rectal resection or abdominoperineal amputation of any etiology.
  * It is a single-center trial.
  * The expected recruitment period is 36 months. The follow-up time of the patients in the study is 30 days.
  * The approximate duration of the study is 3 years.

Calculation of the sample size:

According to published clinical trials, up to 30% of rectal surgery patients who have VS removed will have an AUR for the first POD. The estimated risk of AUR after removal of VS on the 3rd PDO is 5%. If a confidence level at 95% is set and a statistical power of 80% is desired and having an expected proportion of losses of 10% in each group, the sample size should be 48 in each group.

Randomization process:

Patients who meet the inclusion criteria for the study will be randomized using random number generator functions with the SPSS v.25 program in the UC withdrawal group on the first, third and fifth postoperative days. The randomization will be 1: 1: 1.

Allocation concealment will be done by sealed opaque envelopes. The envelope will be opened inside the operating room at the beginning of the surgical procedure.

Masking process:

Patients, surgeons, and research staff know the intervention group to which the patient have been assigned.

Dropouts, withdrawals and losses

* Dropouts: patients included in a clinical trial who are unwilling or unable to continue in the study or in follow-up.
* Withdrawals: patients who are forced to abandon the study due to the appearance of exclusion criteria, but whose follow-up is feasible.
* Loss of follow-up: patients included in the study, who do not carry out the indicated controls, for whom it is not possible to obtain follow-up data.
* Criteria for Inclusion and Exclusion

  • INCLUSION CRITERIA:
* Patients undergoing programmed rectal surgery.
* Age ≥ 18 years and <85 years.
* Any type of tumor, any T, N, M.
* Consent signed by the patient and the researcher.

  • EXCLUSION CRITERIA:
* IPSS> 20
* Transanal resection.
* Urinary catheterization in the 7 days prior to surgery.
* Patients taking treatment for benign prostatic hyperplasia.
* Urine infection in the month prior to surgery.
* Patients with chronic kidney failure with Creatinine> 2 mg / dL.
* Enterovesical fistula.
* Neurogenic bladder.
* Patients with a sacral nerve stimulator or artificial sphincter.
* Inability to read or understand any of the languages of informed consent.
* Emergency surgery.
* Psychiatric illnesses, addictions or any disorder that prevents the understanding of informed consent.
* Description of the intervention:

Management common to all patients included in the study:

Lithotomy position for surgery, regardless of whether it is subsequently modified to the prone position. Laparotomy or laparoscopic surgery, performing Anterior Rectum Resection, Lower Anterior Resection, with or without anastomosis or Abdominoperineal Resection.

Transurethral 16 Fr Foley catheter placement. Balanced general anesthesia, with or without epidural catheter, at the discretion of the responsible anesthesiologist. Avoid hydric overload and favor normothermia.

Positioning of the usual trocars (but modifiable according to the surgeon's preferences). An oncological or transmesorectal mesorectal dissection will be performed according to the needs of each patient, always trying to identify the upper and lower hypogastric plexus, without injuring them. The inferior mesenteric artery will be cut at least 2 cm from the root to avoid the superior hypogastric plexus or a distal ligation with preservation of the left colic artery. The extraction of the sample will be by a Minipfannenstiel, laparotomy or perineum.

In group 1A, the UC will be removed in the first 24 hours after surgery, accompanied by a urine culture taken from UC. In group 1B, the UC will be removed approximately 72 hours after surgery, accompanied by a urine culture taken for UC. In group 1C, the UC will be removed approximately 96 hours after surgery, accompanied by a urine culture taken from UC.

In cases of APR, the UC will be replaced, which will be maintained for at least 4 more days, at which point its removal will be attempted again along with taking another urine culture.

Complications data will be collected together with the other variables in the data collection sheet.

The other fast-track principles approved by different participating centers will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing programmed rectal surgery.
* Age ≥ 18 years and <85 years.
* Any type of tumor, any T, N, M.
* Consent signed by the patient and the researcher.

Exclusion Criteria:

* IPSS> 20
* Transanal local resection.
* Urinary catheterization in the 7 days prior to surgery.
* Patients taking treatment for benign prostatic hyperplasia.
* Urine infection in the month prior to surgery.
* Patients with chronic kidney failure with Creatinine> 2 mg / dL.
* Enterovesical fistula.
* Neurogenic bladder.
* Patients with a sacral nerve stimulator or artificial sphincter.
* Inability to read or understand any of the languages of informed consent.
* Emergency surgery.
* Psychiatric illnesses, addictions or any disorder that prevents the understanding of informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
to compare the incidence of acute urine retention after removal of the urinary catheter in the postoperative period of rectal resection. | 1-30 days
  to compare the incidence of acute urine retention after removal of the urinary catheter in the postoperative period of rectal resection, measured by the proportion of patients that need to be newly catheterized in the first 30 postoperative days.

SECONDARY OUTCOMES:
Incidence of urinary tract infection after urinary catheter removal. | 1-30 days
  Proportion of patients that hace a urinary tract infection measured by the culture obtained at the time of the removal of the catheter.
Incidence of surgical wound infection | 1-30 days
  Incidence of surgical wound infection after rectal resection surgery measured by a positive culture or a drained abscess.
Incidence of respiratory infection | 1-30 days
  Respiratory infection is considered a positive sputum culture and / or a chest radiograph with parenchymal condensations.
Incidence of anastomotic dehiscence | 1-30 days
  The incidence of anastomotic dehiscence and its severity is measured by the International Study Group of Rectal Cancer. Anastomotic dehiscence is defined as a defect of the intestinal wall at the anastomotic site (including suture and staple lines of neorectal reservoirs) leading to a communication between the intra- and extraluminal compartments
Incidence of ileus | 1-30 days
  Incidence of ileus measured by the proportion of patients with delay in oral tolerance due to vomiting, abdominal distension, or the need for nasogastric tube placement.
Incidence of postoperative complications | 1-30 days
  Postoperative complications according to the Comprehensive Complication Index (CCI) scale. The CCI integrates all complications of the Clavien-Dindo classification and offers a metric approach to measure morbidity. Higher rates mean more complications.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Maria Enriquez-Navascues, PhD, Principal Investigator — H Donostia
Locations (1):
- Hospital Donostia, Donostia / San Sebastian, Guipuzcos, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barone JG, Cummings KB. Etiology of acute urinary retention following benign anorectal surgery. Am Surg. 1994 Mar;60(3):210-1. PMID 8116984
- [Background] Sartori CA, Sartori A, Vigna S, Occhipinti R, Baiocchi GL. Urinary and sexual disorders after laparoscopic TME for rectal cancer in males. J Gastrointest Surg. 2011 Apr;15(4):637-43. doi: 10.1007/s11605-011-1459-0. Epub 2011 Feb 17. PMID 21327977
- [Background] Keating JP. Sexual function after rectal excision. ANZ J Surg. 2004 Apr;74(4):248-59. doi: 10.1111/j.1445-2197.2004.02954.x. PMID 15043737
- [Background] George D, Pramil K, Kamalesh NP, Ponnambatheyil S, Kurumboor P. Sexual and urinary dysfunction following laparoscopic total mesorectal excision in male patients: A prospective study. J Minim Access Surg. 2018 Apr-Jun;14(2):111-117. doi: 10.4103/jmas.JMAS_93_17. PMID 28928335
- [Background] Zmora O, Madbouly K, Tulchinsky H, Hussein A, Khaikin M. Urinary bladder catheter drainage following pelvic surgery--is it necessary for that long? Dis Colon Rectum. 2010 Mar;53(3):321-6. doi: 10.1007/DCR.06013e3181c7525c. PMID 20173480
- [Background] Patel DN, Felder SI, Luu M, Daskivich TJ, N Zaghiyan K, Fleshner P. Early Urinary Catheter Removal Following Pelvic Colorectal Surgery: A Prospective, Randomized, Noninferiority Trial. Dis Colon Rectum. 2018 Oct;61(10):1180-1186. doi: 10.1097/DCR.0000000000001206. PMID 30192326
- [Result] Petros JG, Bradley TM. Factors influencing postoperative urinary retention in patients undergoing surgery for benign anorectal disease. Am J Surg. 1990 Apr;159(4):374-6. doi: 10.1016/s0002-9610(05)81274-7. PMID 2316800